CLINICAL TRIAL: NCT04359823
Title: Topical Treatment for Superficial Disseminated Actinic Porokeratosis: A Single-Blinded Comparison Between Lovastatin/Cholesterol and Lovastatin
Brief Title: DSAP Treatment Comparison: 2% Lovastatin/ 2% Cholesterol vs 2% Lovastatin Alone
Acronym: DSAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Dirk Elston, MD, Professor and Chairman, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00096259
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-02

CONDITIONS: Actinic Porokeratosis
MeSH Terms: interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Statin/Cholesterol Combination Group (Experimental): This arm will utilize 2% cholesterol and 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion twice daily for 12 weeks.
  Interventions: Drug: Lovastatin 2%, 2% Cholesterol Cream
- Statin Alone Group (Experimental): This arm will utilize 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion twice daily for 12 weeks.
  Interventions: Drug: Lovastatin 2% Cream

INTERVENTIONS:
Drug: Lovastatin 2%, 2% Cholesterol Cream — Patients selected to the study will be randomly assigned to this arm. They will have a 50% chance of being placed in this arm compared to the other arm.
  Arms: Statin/Cholesterol Combination Group
Drug: Lovastatin 2% Cream — Patients selected to the study will be randomly assigned to this arm. They will have a 50% chance of being placed in this arm compared to the other arm.
  Arms: Statin Alone Group

SUMMARY:
This study will analyze the effects of topical lovastatin/cholesterol vs topical lovastatin alone in patients with disseminated superficial actinic porokeratosis. Patients will be divided into two groups, topical lovastatin/cholesterol and topical lovastatin alone. Patients will apply topical treatment twice daily to lesions over the course of 12 weeks. Follow up will occur in the virtual setting and photographs will be used to document progress.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of cholesterol/lovastatin versus lovastatin alone to treat porokeratosis. Our working hypothesis is that both topical cholesterol/lovastatin and lovastatin alone are helpful in treating patients with disseminated superficial actinic porokeratosis (DSAP). Potential subjects will be approached by their care team member to be made aware of the study at MUSC Dermatology clinics. Subsequently, members of the study team will approach their own patients to ask for participation in this study. Pertinent project information, risks, and time commitment will be relayed to subjects. If subjects show interest in participating, they will be given consent forms to either sign or bring home for consideration. If the patient is eligible for the study, he or she will be randomly assigned to one of two groups. They will have a 50/50 chance of being in either group. You will not make the choice to which group you are assigned. The two groups are Group A (cholesterol/lovastatin) and Group B (lovastatin only). The patient will not be informed of which group they are in and will not be informed of what their study medication is, allowing single-blinding. Researchers will not be masked. Initial enrollment will occur virtually. Enrolled subjects will be followed up at monthly intervals for three months via virtual check-in. At each visit, participants will undergo brief physical examination; additionally, clinical photographs of the lesion will be obtained. Photographs will be stored in the electronic medical record and stored in a departmental secure drive for further analysis of lesion features. At each visit the novel DSAP- General Assessment Scale and RAND36 QoL scale will be administered. Patients will be contacted via virtual check-in visits at weeks 4, 8, and 12. Patients will be asked about compliance and any adverse effects experienced. Participants will also be contacted by phone by study team member to assess for any adverse effects at weeks 2 and 6 of treatment. Compounded topical medication prescribed to subjects will be self-applied twice daily. These medications will be prepared by Tide Water Pharmacy Charleston, SC and Chemistry RX Philadelphia, PA. Chemistry Rx will ship the medications to the patients. They will be prepared so the study will remain single-blinded. The associated costs will not be covered by the research budget. Dermoscopic and clinical photographs will be subsequently analyzed for the presence of cornoid lamella. The team will record any additional dermoscopic or clinicals feature that may arise during the analyses. Frequency of dermoscopic and clinical features will be analyzed against clinical involution to find possible predictors.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years and older with the diagnosis of disseminated superficial actinic porokeratosis.

Exclusion Criteria:

* Patients with allergies or contraindications to lovastatin or cholesterol
* Female patients currently pregnant or lactating.
* Female patients with plans to become pregnant.
* Patients actively taking approved forms of long-term contraception (oral contraceptives, implantable intrauterine devices, or other hormone eluting implants) will be allowed to participate as long as they have no plan to become pregnant during the course of the study. A urine pregnancy test will be administered to these patients to confirm that they can be included in the study.
* Inability or unwillingness of subject or legal guardian/representative to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Elston, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santa Lucia G, Snyder A, Lateef A, Drohan A, Gregoski MJ, Barton V, Elston DM. Safety and Efficacy of Topical Lovastatin Plus Cholesterol Cream vs Topical Lovastatin Cream Alone for the Treatment of Disseminated Superficial Actinic Porokeratosis: A Randomized Clinical Trial. JAMA Dermatol. 2023 May 1;159(5):488-495. doi: 10.1001/jamadermatol.2023.0205. PMID 36947042

RESULTS

PARTICIPANT FLOW:
Groups:
- Statin Alone Group: This arm will utilize 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion twice daily for 12 weeks.
  Lovastatin 2%: Patients selected to the study will be randomly assigned to this arm. They will have a 50% chance of being placed in this arm compared to the other arm.
Period: Overall Study
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Started | 17 | 14
Completed | 17 | 12
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Full Range); unit: years] | 59.2 [40 to 83] | 57.3 [38 to 71] | 58.3 [38 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 4 | 1 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Treatment Efficacy Determined by DSAP-GASI Score (Disseminated Actinic Porokeratosis General Assessment Severity Index)
Description: The primary endpoint was the percentage of lesion clearance after 12 weeks of therapy using an exploratory clinical measure modified from a validated psoriasis index. The Disseminated Actinic Porokeratosis General Assessment Severity Index (DSAP-GASI) included plaque/rim elevation, scaling, and color (0= clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe). Lesions of each patient were graded by 2 blinded physicians before and after treatment.
Time Frame: 12 weeks
Population: Treatment efficacy was based on investigator-standardized patient-documented photographs. Repeat photo documentation was obtained if image quality was inadequate or angle, lighting or location was not standardized to prior photos. Thirty-one subjects enrolled in the study, of which 24 provided clear pictures across all four visits (i.e. ~77%) and were considered in the efficacy analysis.
Measure: Number; unit: Percent decrease in mean DSAP-GASI score
Groups:
- Statin/Cholesterol Combination Group: This arm will utilize 2% cholesterol and 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion daily for 12 weeks.
  Lovastatin 2%, 2% Cholesterol Cream: Patients selected to the study will be randomly assigned to this arm. They will have a 50% chance of being placed in this arm compared to the other arm.
- Statin Alone Group: This arm will utilize 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion daily for 12 weeks.
  Lovastatin 2%: Patients selected to the study will be randomly assigned to this arm. They will have a 50% chance of being placed in this arm compared to the other arm.
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Number analyzed (Participants) | 12 | 12
Percent decrease in mean DSAP-GASI score | 50.0 | 51.4

2. Primary Outcome: Presence of Coronoid Lamella on Dermoscopy (or Photograph).
Description: Dermoscopic and clinical photographs will be subsequently analyzed for the presence of cornoid lamella (well circumscribed, erythematous macule with a peripheral rim of hyperkeratosis). The team will record any additional dermoscopic or clinicals feature that may arise during the analyses.
Time Frame: 12 weeks
Population: unable to complete due to COVID 19 pandemic causing virtual visits for most patients.
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Actinic Keratosis Field Assessment Scale
Description: The Actinic Keratosis Field Assessment Scale measures the percent area covered by actinic keratosis on a scale of 0-4 (0 being 0% and 4 being >50% total area on face or scalp), the severity of hyperkeratosis based upon size of lesion and degree of hyperkeratosis (considered positive findings if >1 actinic keratosis with significant hyperkeratosis and >5mm in diameter), and sun damage severity, measured positive (moderate or severe sun damage) or negative (none or mild damage), based upon severity of erythema, telangiectasia, inflammation, atrophy, and pigmentation disorders. This will be used to determine skin changes (described above) during treatment. A higher score would indicate a worse outcome.
Time Frame: 12 weeks
Population: Unable to accurately assess due to lack of in person visits during the covid 19 pandemic.
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Improvement in Dermatology Quality of Life Index Questionnaire
Description: The patient quality of life scale asks 10 questions gaging how the patient skin condition is currently impacting their life. This questionnaire is a common validated tool, available free online. DLQI interpretation: no effect (0-1), mild effect (2-5), moderate effect (6-10), very large effect (11-20), extreme large effect (21-30). Lower scores represent improved quality of life.
  This was given after every visit at weeks 0, 4, 8, and 12 to access if the cream has contributed to quality of life improvement. The mean difference between the first (week 0) and last score (week 12) was used as the final improvement score.
Time Frame: 12 weeks
Population: 3/31 participants did not return a questionnaire at visit 1 or 4. In the statin group 12/14 returned a questionnaire and 16/17 in the combination group.
Measure: Number; unit: Percent improvement in quality of life
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Number analyzed (Participants) | 16 | 12
Percent improvement in quality of life | 48 | 38

5. Secondary Outcome: Improvement in Overall Appearance of DSAP Lesions
Description: Patients were asked if their overall appearance was better, unchanged, worse. The responses were collected at weeks 4, 8, and 12. Only the final visit (week 12) was used in analysis. Better overall improvement is reported in the data table.
Time Frame: 12 weeks
Population: The numbers in each group do not equal the total number of analyzed participants because some declined to answer.
Measure: Number; unit: participants denoting a score of better
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Number analyzed (Participants) | 15 | 13
participants denoting a score of better | 14 | 12

6. Secondary Outcome: Improvement in Color of DSAP Lesions
Description: Patients were asked if their color was lighter, unchanged, darker. The responses were collected at weeks 4, 8, and 12. Only the final visit (week 12) was used in analysis. Lighter coloring is reported in the data table.
Time Frame: 12 weeks
Population: The numbers in each group do not equal the total number of analyzed participants because some declined to answer.
Measure: Number; unit: participants denoting a score of lighter
Groups:
- Statin Alone Group: This arm will utilize 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion daily for 12 weeks.
  Lovastatin 2% Cream: Patients selected to the study will be randomly assigned to this arm. They will have a 50% chance of being placed in this arm compared to the other arm.
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Number analyzed (Participants) | 15 | 13
participants denoting a score of lighter | 13 | 12

7. Secondary Outcome: Improvement in Size of DSAP Lesions
Description: Patients were asked if their lesion size was smaller, unchanged, or larger. The responses were collected at weeks 4, 8, and 12. Only the final visit (week 12) was used in analysis. The number of participants reporting smaller lesions is reported in the data table.
Time Frame: 12 weeks
Population: The numbers in each group do not equal the total number of analyzed participants because some declined to answer.
Measure: Number; unit: participants denoting smaller size
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
Number analyzed (Participants) | 15 | 13
participants denoting smaller size | 12 | 11

8. Secondary Outcome: Pain and Itch Associated With Treatment
Description: Pain and Itch were measured as increased or decreased at weeks 0, 4, 8, and 12. Week 12 findings reported.
Time Frame: 12 weeks
Population: Two participants did not complete the study from the statin group, thus were not allowed in final analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Statin/Cholesterol Combination Group Itch Decrease; Statin/Cholesterol Combination Group Itch Increase; Statin/Cholesterol Combination Group Pain Decrease; Statin/Cholesterol Combination Group Pain Increase: This arm will utilize 2% cholesterol and 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion daily for 12 weeks.
- Statin Alone Group Itch Decrease; Statin Alone Group Itch Increase; Statin Alone Group Pain Decrease; Statin Alone Group Pain Increase: This arm will utilize 2% lovastatin ointment. It will be compounded by a pharmacist. Ointment will be applied on lesional skin with occlusion daily for 12 weeks.
Arm/Group | Statin/Cholesterol Combination Group Itch Decrease | Statin/Cholesterol Combination Group Itch Increase | Statin Alone Group Itch Decrease | Statin Alone Group Itch Increase | Statin/Cholesterol Combination Group Pain Decrease | Statin/Cholesterol Combination Group Pain Increase | Statin Alone Group Pain Decrease | Statin Alone Group Pain Increase
Number analyzed (Participants) | 17 | 17 | 12 | 12 | 17 | 17 | 12 | 12
Participants | 5 | 1 | 1 | 1 | 2 | 0 | 0 | 0

9. Secondary Outcome: Application Frequency Influence on Disseminated Actinic Porokeratosis General Assessment Severity Index
Description: Measure if applying once or twice a day had an affect on treatment efficacy using the DSAP-GASI described in the primary outcome. Factors included plaque/rim elevation, scaling, and color. (0= clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe). Lower score indicates better outcome.
Time Frame: 12 weeks
Population: Data was analyzed against DSAP-GASI scores that had n=12 for each treatment arm. Frequency was also analyzed in the 24 participants selected for the DSAP-GASI. 8 of those participants happened to be once a day and 16 twice a day.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- DSAP-GASI Score With Once a Day Application: Patients applied either 2% lovastatin alone or 2% Cholesterol/ 2% Lovastatin once a day
- DSAP-GASI Score With Twice a Day Application: Patients applied either 2% lovastatin alone or 2% lovastatin/ 2% cholesterol twice a day.
Arm/Group | DSAP-GASI Score With Once a Day Application | DSAP-GASI Score With Twice a Day Application
Number analyzed (Participants) | 8 | 16
score on a scale | 1.42 [0.77 to 2.06] | 1.54 [0.9 to 2.19]

ADVERSE EVENTS:
Time Frame: 12 weeks per participant (during participants study time period). Cumulatively about 6 months for all participants.
Description: Patients had scheduled visits every 4 weeks and were asked about medication toleration. Participants were also contacted two weeks post/pre appointment about any possible new adverse events or new symptoms.
Arm/Group | Statin/Cholesterol Combination Group | Statin Alone Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 3/17 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Statin/Cholesterol Combination Group (N=17) | Statin Alone Group (N=14)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient noticed a rash on the inside of her right elbow. It was one of the many locations where she applied the cream. The rash has since went away after avoiding application to that area for a few days. She continued to use cream on other areas.
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — Patient emailed and said she "had muscle weakness ( felt like my legs were quivering) after standing in a sailboat to steer for 3 hours under stressful conditions and again after playing 4 hours of croquet in one day". Patient continued with study.
Elevated CK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject's PCP has been monitoring her CK as a result of starting statin therapy. CK 664. PCP recommended continued participation in the study granted significant improvement of DSAP lesions and no symptoms or additional signs relevant to the therapy.

LIMITATIONS AND CAVEATS:
Study was limited by covid pandemic requiring virtual appointments with participants. This prevented study team from acquiring in person dermoscopy data and overall limited physical exam assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT04359823/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT04359823/SAP_001.pdf
  • Informed Consent Form (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT04359823/ICF_002.pdf